CLINICAL TRIAL: NCT05469425
Title: Effect of Home-based Preoperative Exercise Training on Quality of Life After Lung Cancer Surgery: A Randomized Controlled Trial
Brief Title: Home-based Preoperative Exercise Training for Lung Cancer Patients Undergoing Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Pedro Machado, Principal Investigator, Instituto Politécnico de Leiria
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OncoEnergy
Record Dates: First submitted 2022-07-13; First posted 2022-07-21 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Lung Neoplasm
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preoperative home-based exercise training (Experimental): Patients allocated to this group will receive usual care plus a preoperative home-based exercise program consisting of aerobic and resistance exercise. In addition, a physical therapist will carry out weekly telephone supervision with all participants.
  Interventions: Behavioral: Preoperative home-based exercise training
- Control Group (No Intervention): Patients allocated to this group will receive usual care and must complete the outcome measures.
  In addition, a physical therapist will carry out weekly telephone calls with all participants to monitor adverse events.

INTERVENTIONS:
Behavioral: Preoperative home-based exercise training — Home-based aerobic and resistance exercise training (preoperative period)
  Dose of aerobic exercise:
  1. Type: Walking
  2. Frequency: 3 sessions per week
  3. Duration: 30 minutes
  4. Intensity: Rate of perceived exertion on Borg Category Ratio-10 (3-5)
  5. Progression: Increase the walking duration in 10 minutes (after week 2)
  Dose of resistance exercise:
  1. Type: Six exercises for upper and lower limbs using bodyweight and free-wights of 1-2kg
  2. Frequency: 2 sessions per week
  3. Duration: 2 sets x 15 repetitions
  4. Rest in-between sets: 45 seconds
  5. Intensity: Rate of perceived exertion on Borg Category Ratio-10 (3-5)
  6. Progression: Increase the number of sets (3 sets of 15 repetitions after week 2)
  Weekly telephone supervision: A physical therapist will carry out weekly telephone calls with all participants to monitor adverse events and recommend strategies to overcome barriers that arise during the exercise program.
  Arms: Preoperative home-based exercise training

SUMMARY:
Lung cancer accounts for over 11% of global cancer incidence and is the leading cause of cancer death, with numbers in 2020 reaching 1.8 million deaths worldwide.

For early-stage lung cancer patients, surgical resection is the recommended treatment and the intervention associated with a better prognosis. However, in consequence of surgery there is a substantial deterioration in health-related quality of life across most dimensions, especially in the first month, with 100% of lung cancer patients concerned about the limitations in their physical function and 96% about the levels of fatigue and pain after lobectomy.

Additionally, some patients developed postoperative pulmonary complications, which are associated with increased length of hospital stay and higher risk of mortality.

In this context, and considering that the number of lung cancer cases with an indication for surgery will increase by 60% from 2018 to 2040, to find feasible and effective interventions that could optimize postoperative recovery is of major clinical relevance.

The primary purpose of this study will be to evaluate the efficacy of home-based preoperative exercise training to improve health-related quality of life after lung cancer surgery. The secondary purpose of this study will be to evaluate the efficacy of the home-based exercise program to improve physical performance and to reduce postoperative complications /length of hospital stay. Participants will be randomly allocated to a preoperative exercise intervention, that will consist of combined aerobic and resistance exercise, or to a control group that will receive usual care (i.e., no exercise training).

Based on the strong evidence indicating a therapeutic effect of exercise training on fatigue and physical function, domains of HRQOL especially affected after lung cancer surgery, the investigators hypothesized that the home-based exercise program will be effective to improve these domains before surgery and attenuate its deterioration after surgery, optimizing the recovery in postoperative HRQOL.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for surgical treatment of suspected or confirmed lung cancer (clinical stage IIIA or less)
* Waiting time for surgery of at least two weeks from baseline assessment
* Medical clearance to exercise.
* Signed informed consent prior to initiation of study-related procedures

Exclusion Criteria:

* Metastatic cancer
* Presence of physical or mental disabilities that contraindicated exercise training or physical testing
* Unable to communicate in Portuguese or English
* Performing combined aerobic plus resistance training over the past month (self-reported ≥2 days a week, ≥30 minutes each session).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Changes in health-related quality of life | Baseline to 2-3 days before surgery
  Will be assessed through the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) (version 3.0). The QLQ-C30 is composed of 30 questions, including five multi-item functioning scales, three multi-item symptom scales, six single-item symptom scales, and a two-item global health status scale [GHS]. Scores range from 0 to 100 points, with a higher score on the functioning scales indicating a higher level of functioning, whereas a higher score on the symptom scales indicates a higher level of symptom burden.
  In addition, the investigators will assess EORTC QLQ-C30 summary score (SumSc) because it provides a psychometrically more robust alternative to the GHS score that is frequently used as the primary HRQOL endpoint in clinical trials. The SumSc is calculated from the mean of 13 of the 15 QLQ-C30 scores (the GHS and financial impact scales are excluded).
Changes in health-related quality of life | Baseline to 3-5 weeks after surgery
  Will be assessed through the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire C30 (QLQ-C30) (version 3.0). The QLQ-C30 is composed of 30 questions, including five multi-item functioning scales, three multi-item symptom scales, six single-item symptom scales, and a two-item global health status scale [GHS]. Scores range from 0 to 100 points, with a higher score on the functioning scales indicating a higher level of functioning, whereas a higher score on the symptom scales indicates a higher level of symptom burden.
  In addition, the investigators will assess EORTC QLQ-C30 summary score (SumSc) because it provides a psychometrically more robust alternative to the GHS score that is frequently used as the primary HRQOL endpoint in clinical trials. The SumSc is calculated from the mean of 13 of the 15 QLQ-C30 scores (the GHS and financial impact scales are excluded).

SECONDARY OUTCOMES:
Changes in exercise capacity | Baseline to 2-3 days before surgery
  Will be assessed by the Incremental Shuttle Walk Test (ISWT). The ISWT measures the distance in meters an individual can walk around a 10 meters shuttle course paced according to an incremental speed dictated by an audio recording and was performed under the supervision of a single investigator using the protocol described by Singh et al. (1992). The test finished when the participant can no longer maintain the desired speed or became too breathless to continue.
Changes in exercise capacity | Baseline to 3-5 weeks after surgery
  Will be assessed by the Incremental Shuttle Walk Test (ISWT). The ISWT measures the distance in meters an individual can walk around a 10 meters shuttle course paced according to an incremental speed dictated by an audio recording and was performed under the supervision of a single investigator using the protocol described by Singh et al. (1992). The test finished when the participant can no longer maintain the desired speed or became too breathless to continue.
Changes in handgrip strength | Baseline to 2-3 days before surgery
  Will be assessed using the Hamar plus+ digital hand dynamometer. Measurements will be conducted using the standard position approved by the American Society of Hand Therapists. The standard adjustable handle dynamometer will be set at the second handle position for all patients. The non-tested arm will be resting neutrally and both feet were firmly on the ground, shoulder width apart. Patients will be instructed to grip the handle with maximal strength during 3 seconds and the measurements will be repeated three times for the left and right hand, with 30 seconds rest in-between measurements. The highest value for both hands (in kilograms) will be considered as the output measure to each patient.
Changes in handgrip strength | Baseline to 3-5 weeks after surgery
  Will be assessed using the Hamar plus+ digital hand dynamometer. Measurements will be conducted using the standard position approved by the American Society of Hand Therapists. The standard adjustable handle dynamometer will be set at the second handle position for all patients. The non-tested arm will be resting neutrally and both feet were firmly on the ground, shoulder width apart. Patients will be instructed to grip the handle with maximal strength during 3 seconds and the measurements will be repeated three times for the left and right hand, with 30 seconds rest in-between measurements. The highest value for both hands (in kilograms) will be considered as the output measure to each patient.
Changes in five times sit to stand test | Baseline to 2-3 days before surgery
  Patients will be instructed to perform the Five Times Sit to Stand Test (5STS) on a standardized armless chair (i.e., seating height between 41-45 cm, no elbow rests and wheels). After the cue "ready, set, go!", patients will start the STS repetitions as rapidly as possible from the sitting position with their buttocks touching the chair to the full standing position, with their arms crossed over the chest. The 5STS test will finish when the patients sit on the chair after the fifth repetition, and the time needed to complete the task will be recorded with a stopwatch to the nearest 0.01 s.
Changes in five times sit to stand test | Baseline to 3-5 weeks after surgery
  Patients will be instructed to perform the Five Times Sit to Stand Test (5STS) on a standardized armless chair (i.e., seating height between 41-45 cm, no elbow rests and wheels). After the cue "ready, set, go!", patients will start the STS repetitions as rapidly as possible from the sitting position with their buttocks touching the chair to the full standing position, with their arms crossed over the chest. The 5STS test will finish when the patients sit on the chair after the fifth repetition, and the time needed to complete the task will be recorded with a stopwatch to the nearest 0.01 s.
Postoperative length of hospital stay | 3-6 days after surgery
  Defined as the number of days patients spend in the hospital after surgery. This will be collected from individual clinical records.
Postoperative complications | 30 days after surgery
  Will be assessed using the Comprehensive Complication Index, that integrates all complications with their respective severities on a continuous scale ranging from 0 (no burden due to complications) to 100 (death as a result of complications).Postoperative complications were scored by severity using the scored by severity using the Clavien-Dindo classification.
Adverse events | Baseline to 2-3 days before surgery
  Defined as any unfavorable or unexpected event that occurred as a direct result of exercise training, during or within 24 hours after an exercise session. The severity of adverse events will be categorized based on the Common Terminology Criteria for Adverse Events (CTCAE), version 5. The CTCAE provides a grading (severity) scale, with each adverse event been classified as grade 1 (asymptomatic or mild symptoms, clinical or diagnostic observations only, and/or intervention not indicated) to grade 5 (death). An adverse event will be classified as "serious" if it resulted in hospitalization, persistent or significant disability, was life threatening, or resulted in death (i.e., grade 3 or higher).
Exercise attendance rate | Baseline to 2-3 days before surgery
  Attendance rate will be defined as the ratio of total completed to planned exercise sessions, expressed as a percentage.
Exercise compliance rate | Baseline to 2-3 days before surgery
  Compliance rate will be defined as the ratio of total completed to planned training volume, expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro FA Machado, Principal Investigator — Center for Innovative Care and Health Technology, Polytechnic of Leiria
Locations (1):
- Portuguese Oncology Institute of Coimbra, Coimbra, Portugal